CLINICAL TRIAL: NCT06689631
Title: Efficacy of Mucociliary Clearance Techniques in Non-hospitalised Infants with Acute Bronchiolitis
Brief Title: Mucociliary Clearance Techniques for Acute Bronchiolitis
Acronym: CLEARBRONCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Raquel Leirós-Rodríguez, Principal investigator and Associate Professor, Universidad de León
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETICA-ULE-062-2023; ULE (Other: Universidad de León)
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Bronchiolitis Due to Respiratory Syncytial Virus; Bronchiolitis Acute; Bronchiolitis Acute Viral
Keywords: mucociliary clearance; respiratory physiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): The intervention consisted of a Respiratory Physiotherapy session including: mucociliary clearance techniques (prolonged slow expiration and provoked cough), bronchodilator when prescribed and nebulisation with 3% hypertonic saline.
  Interventions: Procedure: Respiratory Physiotherapy

INTERVENTIONS:
Procedure: Respiratory Physiotherapy — Mucociliary clearance techniques (prolonged slow expiration and provoked cough), bronchodilator when prescribed and nebulisation with 3% hypertonic saline.

SUMMARY:
To assess the efficacy of mucociliary clearance techniques in non-hospitalised infants with a first episode of mild to moderate acute bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of first episode of acute Bronchiolitis.
* Acute Bronchiolitis with mild (ESBA score = 1-4) or moderate (ESBA score =5-9) severity according to the ESBA.
* Informed consent signed by parents or legal guardians.

Exclusion Criteria:

* Infants previously diagnosed with chronic respiratory disease.
* Previous episodes of wheezing.
* Presence of any type of contraindication to receive Respiratory Physiotherapy treatment.

Ages: 28 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
ESBA | 1 session (45 minutes)
  The variables collected using the ESBA scale were: wheezing, crackles, inspiratory effort, Inspiratory/Expiratory ratio, respiratory rate and heart rate.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez Bellido V, Velaz Baza V, Esteo MDCJ, Carballo RG, Colombo A, Zaldivar JNC, Donadio MVF. Safety of airway clearance combined with bronchodilator and hypertonic saline in non-hospitalized infants with acute bronchiolitis. Arch Pediatr. 2021 Nov;28(8):707-711. doi: 10.1016/j.arcped.2021.09.007. Epub 2021 Oct 5. PMID 34625378